CLINICAL TRIAL: NCT00140556
Title: Concurrent Angiogenic and EGFR Blockade in Conjunction With Curative Intent Chemoradiation for Locally Advanced Head and Neck Cancer
Brief Title: Angiogenic and EGFR Blockade With Curative Chemoradiation for Advanced Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: David M. Brizel, MD (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, David M. Brizel, MD, Professor, Radiation Oncology, Duke University
Organization: Duke University (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008840; 7077 (Other: Legacy IRB number)
Record Dates: First submitted 2005-08-29; First posted 2005-09-01 (Estimated); Results first posted 2011-08-31 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Head and Neck Cancer; Pharynx Cancer
Keywords: head and neck cancer; targeted therapy; bevacizumab; erlotinib; Tarceva; radiotherapy; concurrent chemotherapy; pharynx cancer; tonsil cancer; hyperfractionation; angiogenesis; epidermal growth factor; vascular endothelial growth factor; magnetic resonance spectroscopy; cancer of the head and neck; upper aerodigestive tract neoplasms; pharynx neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms; Pharyngeal Neoplasms; Tonsillar Neoplasms | interventions — Chemoradiotherapy; Cisplatin; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ChemoRadiotherapy (Experimental): Radiation Therapy concurrent with cisplatin chemotherapy, Avastin and Tarceva
  Interventions: Radiation: Chemoradiotherapy; Drug: Cisplatin; Drug: Bevacizumab; Drug: Erlotinib

INTERVENTIONS:
Radiation: Chemoradiotherapy — External beam radiation daily (M-F)
Drug: Cisplatin — Cisplatin week 1 and 5 of radiation
Drug: Bevacizumab — Bevacizumab (Avastin) day 1 of weeks 1, 3, and 5 of radiation
  Other Names: Avastin
Drug: Erlotinib — Erlotinib daily during radiation
  Other Names: Tarceva

SUMMARY:
Radiotherapy (RT) with concurrent chemotherapy represents the state of the art in curative intent treatment for locally advanced squamous carcinoma of the head and neck. Tumor hypoxia and high levels of angiogenesis (blood vessel formation) are associated with treatment failure. Preclinical models reveal that radiotherapy itself may induce tumor secretion of vascular endothelial growth factor (VEGF). Curability may consequently be reduced by multiple mechanisms. Over-expression of epidermal growth factor receptor (EGFR) also occurs commonly and increases the risk of treatment failure. The addition of EGFR blockade to RT alone increases the chance of a cure. Concurrent VEGF and EGFR blockade could be synergistic with one another and improve the effectiveness of concurrent chemoradiation for advanced head and neck cancer.

This study will add angiogenic and epidermal growth factor receptor (EGFR) blockade into an established program of curative intent concurrent chemoradiation for locally advanced head and neck cancer. The safety and effectiveness of delivering the drugs bevacizumab and Tarceva in conjunction with twice daily irradiation and concurrent cisplatin (CDDP) chemotherapy will be determined.

DETAILED DESCRIPTION:
Pre Radiation Period:

* Bevacizumab (10 mg/kg) on days -14 and 0, or
* Tarceva (100 mg) daily from -14-0, or
* Bevacizumab (10 mg/kg) on days -14 and 0; Tarceva (100 mg) daily from -14-0

Chemoradiation Period:

* Radiotherapy may be delivered via conventional 2-D, conformal 3-D, or intensity modulated (IMRT) technique as is clinically indicated. Radiotherapy and CDDP doses will be delivered uniformly to all treatment cohorts:

  * RT: 1.25 Gy BID M-F with a 6 hour interfraction interval
  * Treatment break during week 4. Total dose 70 Gy/7 weeks
  * CDDP: 33 mg/m2 M-W on weeks 1 and 5 of RT with standard DUMC hydration and anti-emetic regimens
* Bevacizumab (10mg/kg): Monday of weeks 1, 3, 5, 7 of RT
* Tarceva (100 mg): Daily for weeks 1-7 of treatment, except for days receiving CDDP

Safety Assessments:

* Baseline and then weekly assessments of blood pressure and urine protein : creatinine ratios during lead in and chemoRT phases of treatment
* Baseline carotid Doppler ultrasound evaluation
* Carotid Doppler ultrasound evaluation 1 month post-chemoRT

Efficacy Assessments:

* MR Imaging/Spectroscopy to be done at baseline, end of lead-in phase, end of week 1 of chemoRT, and end of chemoRT
* Angiogenic and EGFR related cytokines. Specifically, blood samples will be obtained to assay levels of VEGF, b-FGF, IL-8, D-dimer, EGF, TGF. These samples will be obtained on the same dates as the MR studies with an additional set of samples obtained at the midpoint of the lead in phase of treatment (day -7).

Clinical Assessments:

* All patients will undergo a minimum of once weekly interval history and physical examination including fiberoptic pharyngoscopy/laryngoscopy when indicated in the Department of Radiation Oncology to monitor for side effects and response to treatment as per standard routine for the care of patients with head and neck cancer.
* Patient compliance with Tarceva administration monitored via diary MRI/MRS (Magnetic Resonance Spectroscopy) DE-MRI

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced squamous carcinoma of the head and neck (AJCC stages II/IV, M0, and excluding T1N1 and T1N2) undergoing curative intent concurrent chemoradiation.
* Previous treatment of any sort other than a biopsy is not allowed.
* Eligible anatomic sites:

  * oral cavity
  * oropharynx
  * hypopharynx
  * supraglottic
  * glottic larynx
* KPS > 60

Exclusion Criteria:

* Nasopharynx primary
* History of malignancy other than basal cell skin cancer.
* History of claudication, bleeding, or thromboembolic disorders. Patients receiving heparin or Coumadin therapy are ineligible.
* Primary tumor or lymph node encasement of the carotid artery
* Blood pressure of >150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0; anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations, or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein : creatinine ratio ≥ 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* AST, ALT, or bilirubin > 1.5 x normal
* PT or PTT > 1.5 x normal
* Platelets < 100,000
* WBC < 2000
* Hgb < 10
* Creatinine clearance < 60 mL/hr
* Refusal to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-08; Primary Completion 2009-05 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brizel, MD, Principal Investigator — Department of Radiation Oncology; Duke University Medical Center
Locations (1):
- Department of Radiation Oncology; Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Brizel DM, Dodge RK, Clough RW, Dewhirst MW. Oxygenation of head and neck cancer: changes during radiotherapy and impact on treatment outcome. Radiother Oncol. 1999 Nov;53(2):113-7. doi: 10.1016/s0167-8140(99)00102-4. PMID 10665787
- [Background] Brizel DM, Albers ME, Fisher SR, Scher RL, Richtsmeier WJ, Hars V, George SL, Huang AT, Prosnitz LR. Hyperfractionated irradiation with or without concurrent chemotherapy for locally advanced head and neck cancer. N Engl J Med. 1998 Jun 18;338(25):1798-804. doi: 10.1056/NEJM199806183382503. PMID 9632446
- [Background] Brizel DM, Schroeder T, Scher RL, Walenta S, Clough RW, Dewhirst MW, Mueller-Klieser W. Elevated tumor lactate concentrations predict for an increased risk of metastases in head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Oct 1;51(2):349-53. doi: 10.1016/s0360-3016(01)01630-3. PMID 11567808
- [Background] Dewhirst MW, Poulson JM, Yu D, Sanders L, Lora-Michiels M, Vujaskovic Z, Jones EL, Samulski TV, Powers BE, Brizel DM, Prosnitz LR, Charles HC. Relation between pO2, 31P magnetic resonance spectroscopy parameters and treatment outcome in patients with high-grade soft tissue sarcomas treated with thermoradiotherapy. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):480-91. doi: 10.1016/j.ijrobp.2004.06.211. PMID 15667971
- [Background] Moeller BJ, Cao Y, Li CY, Dewhirst MW. Radiation activates HIF-1 to regulate vascular radiosensitivity in tumors: role of reoxygenation, free radicals, and stress granules. Cancer Cell. 2004 May;5(5):429-41. doi: 10.1016/s1535-6108(04)00115-1. PMID 15144951
- [Result] Craciunescu O, Brizel D, Cleland E, Yoo D, Muradyan N, Carroll M, Barboriak D, MacFall J. Dynamic contrast enhanced-MRI in head and neck cancer patients: variability of the precontrast longitudinal relaxation time (T10). Med Phys. 2010 Jun;37(6):2683-92. doi: 10.1118/1.3427487. PMID 20632579
- [Derived] Yoo DS, Kirkpatrick JP, Craciunescu O, Broadwater G, Peterson BL, Carroll MD, Clough R, MacFall JR, Hoang J, Scher RL, Esclamado RM, Dunphy FR, Ready NE, Brizel DM. Prospective trial of synchronous bevacizumab, erlotinib, and concurrent chemoradiation in locally advanced head and neck cancer. Clin Cancer Res. 2012 Mar 1;18(5):1404-14. doi: 10.1158/1078-0432.CCR-11-1982. Epub 2012 Jan 17. PMID 22253412
- [Derived] Craciunescu OI, Yoo DS, Cleland E, Muradyan N, Carroll MD, MacFall JR, Barboriak DP, Brizel DM. Dynamic contrast-enhanced MRI in head-and-neck cancer: the impact of region of interest selection on the intra- and interpatient variability of pharmacokinetic parameters. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):e345-50. doi: 10.1016/j.ijrobp.2011.05.059. Epub 2011 Oct 8. PMID 21985945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the multidisciplinary ENT or Radiation Oncology Clinics between September 2005 and February 2009.
Period: Pre Radiation Period: Avastin / Tarceva
Arm/Group | Entire Study Population
Started | 28
Completed | 28
Not Completed | 0
Period: Chemoradiotherapy Period
Arm/Group | Entire Study Population
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 28
Feeding Tube [Number; unit: Participants] — Feeding tube present before start of treatment
  Participants
    Feeding Tube Present Baseline | 4
    No Feeding Tube at Baseline | 24

OUTCOME MEASURES:

1. Primary Outcome: Tumor Resolution
Description: Complete response (resolution) of tumor on clinical exam.
Time Frame: Within 30 days of completing RT
Population: 2 participants had occult primaries, thus were not included in clinical complete response
Measure: Number; unit: Participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 26
Participants | 25

2. Secondary Outcome: Local Regional Control
Time Frame: 1 yr following chemoradiation
Reporting Status: Not Posted

3. Secondary Outcome: Failure Free Survival
Time Frame: 3 yrs
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Acute adverse events through 30 days post end of treatment. Possibly related to chemoradiotherapy greater than grade 1. Late radiotherapy related adverse events through 2 years.
Description: Toxicity assessment weekly during treatment, and post treatment at 1 month and every 3 months through year 2.
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 15/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=28)
Bradycardia (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 7 (7)
Febrile Neutropenia (Infections and infestations) | 3 (4)
Fever (General disorders) | 3 (3) — Fever (in the absence of neutropenia)
Mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=28)
Anorexia (Gastrointestinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 18
Dental, periodontal disease (Gastrointestinal disorders) | 3 (3) — Late radiation effect
Diarrhea (Gastrointestinal disorders) | 5
Dry Mouth (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 9
Hiccough (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Cardiac disorders) | 4
Mucosal Infection (Infections and infestations) | 17 — Oral candiasis
Mucositis, Oropharyngeal (Gastrointestinal disorders) | 26
Nausea (Gastrointestinal disorders) | 21
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 (5) — Late radiation effect
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 15 — Erlotinib (Tarceva) rash
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 3 (3) — Late radiation effect
Vomiting (Gastrointestinal disorders) | 8
Weight Loss (General disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less